CLINICAL TRIAL: NCT02943265
Title: Care Coordination for Complex Cancer Survivors in an Integrated Safety Net System (Project Connect)
Brief Title: Care Coordination for Complex Cancer Survivors in an Integrated Safety Net System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Simon Craddock Lee, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STU 102015-090
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Colorectal Cancer
Keywords: Care Coordination
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complex Care Survivors (Experimental): Patients eligible for the study who will receive Care Coordination Strategies.
  Interventions: Other: Care Coordination Strategies

INTERVENTIONS:
Other: Care Coordination Strategies — Co-located Care coordinator will use EMR-driven registry to facilitate patient transitions between primary care and oncology care and enhance teamwork through coaching and technical assistance.

SUMMARY:
Nearly 70% of people living with cancer are "complex patients" with multiple chronic conditions who must deal not only with effects of their cancer but also continuing diseases such as diabetes, depression, hypertension, or heart disease. Care coordination strategies shown to be effective in improving outcomes for common medical conditions seen in primary care include: systematic transitions for patients to and from specialty care; intensive case management; and a team-based approach to comprehensive care. Despite an Institute of Medicine report suggesting these strategies as potential ways to improve care for cancer survivors, their implementation has not yet been evaluated for cancer survivors. Parkland Health and Hospital Systems will be implementing care coordinator strategies as part of as quality assurance/quality improvement activities, which Aim 2 and Aim 3 (research components) will evaluate. This protocol has been organized to reflect this distinction between the aims. The investigators expect no more than 1500 patients to be included in these study aims.

DETAILED DESCRIPTION:
This project is a pragmatic trial. The investigators propose a quasi-experimental design where data will be collected both pre- and post-intervention on distinct cross-sections of patients with one or more highly prevalent ambulatory-sensitive chronic conditions (diabetes, hypertension, chronic lung disease, chronic kidney disease, depression, or heart disease) and newly diagnosed with breast, colorectal, or gynecologic cancers (complex cancer survivors) in the Parkland Health & Hospital system (Dallas, TX).

Guided by the "Primary Care Change Model", Parkland will implement evidence-based care coordination strategies to improve care for complex cancer survivors in this integrated safety-net system as a part of quality assurance/quality improvement activities (Aim 1), then this study will comprehensively evaluate how these strategies are implemented in the safety-net setting (Aim 3), and whether implementing these strategies improves care coordination and care outcomes (Aim 2) within the Parkland Health and Hospital System. Investigators expect approximately 1000 new survivors with ≥ 1 prevalent chronic condition to be eligible. The project does not include patients diagnosed with in situ and metastatic disease (Stages 0 and IV) due to insufficient evidence for routine follow-up and management; many of the latter continue indefinitely on active treatment for symptom management. The chronic conditions selected for inclusion are the most prevalent conditions cancer survivors have at Parkland as well as nationally.

* Aim 1: (Quality Assurance/ Improvement) Implement a system-level EMR-driven intervention for approximately 1000 complex cancer survivors at Parkland, combining three evidence-based care coordination strategies; (1) EMR-driven registry to facilitate patient transitions between primary care and oncology care, (2) co-locate a nurse practitioner trained in care coordination within a complex care team, and (3) enhance teamwork through coaching and technical assistance;
* Aim 2: (Research component) Test effectiveness of the strategies on system- and patient-level outcomes using a rigorous, quasi-experimental design with outcomes measured before and after implementation;
* Aim 3: (Research Component) Elucidate system and patient factors that facilitate or hinder implementation and result in differences in experiences of care coordination between complex patients with and without cancer. Investigators will collect quantitative (EMR data, patient surveys) and qualitative (structured observations, patient and provider interviews, EMR audits) data throughout.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over 18 years of age;
2. AND diagnosed with Stage I-III incident breast or colorectal cancers;
3. AND with one or more of the following highly prevalent ambulatory-sensitive chronic conditions (diabetes, hypertension, chronic lung disease, chronic kidney disease, depression, or heart disease).

Exclusion Criteria:

1. Patients with in situ cancers (Stage 0) and those with metastatic disease (Stage IV);
2. OR Patients with impaired hearing or speech;
3. OR Inability to speak English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4322 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Craddock Lee, PhD, MPH, Principal Investigator — University of Texas Southwestern Medical Center; Bijal Balasubramanian, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center Department of Population and Data Sciences, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SJC, Jetelina KK, Marks E, Shaw E, Oeffinger K, Cohen D, Santini NO, Cox JV, Balasubramanian BA. Care coordination for complex cancer survivors in an integrated safety-net system: a study protocol. BMC Cancer. 2018 Dec 4;18(1):1204. doi: 10.1186/s12885-018-5118-7. PMID 30514267

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Parkland Health and Hospital System in Dallas, Texas, USA from September 2017 - April 2021 with all follow up complete by April 30, 2022.
  A retrospective comparison group was derived from Electronic Health Record (EHR) data.
Groups:
- Project CONNECT Care Coordination: Patients with a primary diagnosis of stage I-III breast or colorectal cancer between September 1, 2017, and April 31, 2021 and a diagnosis of at least one comorbid chronic conditions (diabetes, hypertension, heart disease, chronic kidney disease, and chronic obstructive pulmonary disease). Eligible patients received care coordination strategies to facilitate patient transitions between primary care and oncology care.
- Retrospective Comparison Group: Patients with a primary diagnosis of stage I-III breast or colorectal cancer between January 1, 2010 - December 31, 2016 and a diagnosis of at least one comorbid chronic conditions (diabetes, hypertension, heart disease, chronic kidney disease, and chronic obstructive pulmonary disease).The retrospective cohort serves as a comparison group to the care coordination cohort.
- Non-Cancer Retrospective Group: A random sample of 1,000 patients seen January 1, 2010-December 31, 2016 with no history of cancer, at least two chronic conditions (diabetes, hypertension, chronic lung dis-ease, chronic kidney disease, or heart disease). This arm is used as a control to the retrospective comparison group.
Period: Overall Study
Arm/Group | Project CONNECT Care Coordination | Retrospective Comparison Group | Non-Cancer Retrospective Group
Started | 648 | 2674 | 1000
Eligible After Review (Initial eligibility based on EHR data extraction. A detailed review by study team was conducted to confirm all eligibility criteria met.) | 634 | 2092 | 1000
Completed | 634 | 2092 | 1000
Not Completed | 14 | 582 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-Cancer Retrospective Group: A random sample of 1,000 patients seen January 1, 2010-December 31, 2016 with no history of cancer, at least two chronic conditions (diabetes, hypertension, chronic lung dis-ease, chronic kidney disease, or heart disease). This arm is used as a control to the retrospective cancer group.
- Total: Total of all reporting groups
Arm/Group | Project CONNECT Care Coordination | Retrospective Comparison Group | Non-Cancer Retrospective Group | Total
Number analyzed (Participants) | 634 | 2092 | 1000 | 3726
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (14.8) | 54.6 (11.6) | 52.8 (12.9) | 54.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 498 | 1687 | 544 | 2729
  Male | 136 | 405 | 456 | 997
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 285 | 851 | 461 | 1597
  Not Hispanic or Latino | 345 | 1241 | 539 | 2125
  Unknown or Not Reported | 4 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 0 | 3
  Asian | 25 | 101 | 17 | 143
  Native Hawaiian or Other Pacific Islander | 4 | 7 | 0 | 11
  Black or African American | 234 | 736 | 375 | 1345
  White | 363 | 1224 | 597 | 2184
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 8 | 19 | 11 | 38

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Complex Cancer Survivors Meeting Quality of Care Guidelines for Chronic Conditions and Follow-up Cancer Surveillance
Description: Proportion of complex cancer survivors meeting quality of care guidelines for multiple chronic conditions and follow-up cancer surveillance
Time Frame: 5 years
Population: COVID pandemic prevented community health system from being able to extract these data within study timeframe which prevented reporting and analysis on this outcome.
Arm/Group | Project CONNECT Care Coordination | Retrospective Comparison Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Patient Perception of Care (Scale)
Description: Patient-reported perception of care coordination was measured using the Coordination of Care dimension adapted from the validated Picker Patient Experience Questionnaire. The adapted version used in this study consisted of eight items and was administered at baseline and at 6 and 12-months of follow-up. Each item is weighted from 1 to 3 and the cumulative care coordination score is the summation of all the survey items on a scale of 8 to 24. A Lower score indicates better care coordination.
Time Frame: Administered at baseline, 6, and 12 months
Population: This analysis included participants who completed at least one assessment with all care coordination items completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Project CONNECT Care Coordination: Patients with a primary diagnosis of stage I-III breast or colorectal cancer between September 1, 2017, and April 31, 2021 and a diagnosis of at least one of the comorbid chronic conditions (diabetes, hypertension, heart disease, chronic kidney disease, and chronic obstructive pulmonary disease). Eligible patients received care coordination strategies.
Arm/Group | Project CONNECT Care Coordination
Number analyzed (Participants) | 294
score on a scale
  Baseline Survey: number analyzed (Participants) | 241
  Baseline Survey | 11.4 (2.71)
  6-Month Survey: number analyzed (Participants) | 179
  6-Month Survey | 11.2 (2.37)
  12-Month Survey: number analyzed (Participants) | 111
  12-Month Survey | 10.8 (2.26)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time a patient was considered eligible through the final assessment (12 months after enrollment).
Description: Patients in the Retrospective Comparison group and Non-Cancer Historical Group were derived through EHR data extraction with no direct engagement with the study team. Adverse Events were not monitored/assessed for participants from these groups.
Arm/Group | Project CONNECT Care Coordination | Retrospective Comparison Group | Non-Cancer Retrospective Group
All-Cause Mortality (participants affected / at risk) | 39/634 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 39/634 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/634 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Project CONNECT Care Coordination (N=634) | Retrospective Comparison Group (N=0) | Non-Cancer Retrospective Group (N=0)
Participant Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 39 (39) | NA | NA

LIMITATIONS AND CAVEATS:
Survey accrual was lower than target (N=402). Revised power calculations for the analysis of the patient-level primary outcome measure, change in patient perception of care coordination, demonstrated the actual survey sample (N=294) was large enough to detect meaningful improvement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT02943265/Prot_SAP_000.pdf